CLINICAL TRIAL: NCT04601363
Title: Personalized Spine Study Group (PSSG) Registry of Patients With Personalized Spine Rod Implantation
Brief Title: Personalized Spine Study Group (PSSG) Registry
Acronym: PSSG
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Personalized Spine Study Group (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20-2016
Record Dates: First submitted 2020-09-28; First posted 2020-10-23 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Scoliosis; Adolescence; Degenerative Disc Disease; Spinal Fusion; Kyphoscoliosis; Pseudoarthrosis of Spine; Spinal Stenosis; Kyphoses, Scheuermann
MeSH Terms: conditions — Scoliosis; Intervertebral Disc Degeneration; Spinal Stenosis; Scheuermann Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Personalized SpineRods: The patient is being treated with the patient-specific rod with a surgery date planned
  Interventions: Device: Patient Specific Rod
- Patient with other hardware: Patients with other hardware not patient-specific

INTERVENTIONS:
Device: Patient Specific Rod — Posterior spinal fusion rod
  Groups: Patients with Personalized SpineRods

SUMMARY:
The primary objective of the study is a data collection initiative. The study will collect clinical and radiographic outcomes of patients implanted with patient specific rods. The secondary objective is to collect clinical and radiographic outcomes of patients with hardware as a control cohort to the patient-specific rods.

DETAILED DESCRIPTION:
The registry follows patient during their standard of care visits. During a standard of care visit, a study subject will be required to answer questions about themselves and fill out patient reported outcome questionnaires. Spinopelvic measurements will be collect from standard of care x-rays. This registry is observational only used to address patient outcomes sagittal profile through the pre-operative, plan and post-operative events. Rod effectiveness in conjunction with other surgical implants by fusion assessment and sagittal alignment measurements. Patient outcomes in subgroups defined by surgery performed, comorbidities, radiographic measurement, or other outcome variables. Rod curvature maintenance during the follow-up period. Better understanding of the post-operative risks and complications from the pre-operative condition.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been/ will be operated and instrumented with patient-specific rod or spine hardware (control cohort)
* Patient able to consent or assent

Exclusion Criteria:

* Patient unable to sign an informed consent form
* Patient unable to complete a self-administered questionnaire
* Patient is pregnant or planning on becoming pregnant during the duration of their study participation
* Patient is older than 85
* Patient is younger than 10

Ages: 10 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population is implanted with either spine hardware or is undergoing surgery to have patient-specific rod implanted
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-10-29 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Patient-Specific Hardware Spino-Pelvic Measurements | Up to 4 years
  The study will collect clinical and radiographic outcomes of patients implanted with patient specific rods. Measurements are collected from the inferior endplate of the vertebral body C2 to the superior endplate of vertebral body S1 on the lateral view x-ray and from the superior endplate of vertebral body T1 to the superior endplate of vertebral body S1 in the Anteroposterior view x-ray.

SECONDARY OUTCOMES:
Non Patient-Specific Hardware Spino-Pelvic Measurements | 1 year
  The study will collect clinical and radiographic outcomes of patients implanted rods. Measurements are collected from the inferior endplate of the vertebral body C2 to the superior endplate of vertebral body S1 on the lateral view x-ray and from the superior endplate of vertebral body T1 to the superior endplate of vertebral body S1 in the Anteroposterior view x-ray.

OTHER OUTCOMES:
PROMIS CAT Physical Function | Up to 4 years
  Questionnaire regarding physical function of subject
PROMIS CAT Pain | Up to 4 years
  Questionnaire regarding pain of subject
PROMIS CAT Anxiety | Up to 4 years
  Questionnaire regarding anxiety of subject
PROMIS CAT Depression | Up to 4 years
  Questionnaire regarding depression of subject
PROMIS CAT Satisfaction Activity Roles | Up to 4 years
  Questionnaire regarding normal daily activity of subject
Oswestry Disability Index questionnaire (thoracic, thorocolumbar, lumbar surgery) | Up to 4 years
  Oswestry Disability Index questionnaire regarding levels of disability of subject
Neck Disability Index questionnaire (Neck surgery only) | Up to 4 years
  Neck Disability Index questionnaire regarding levels of neck disability of subject
Visual analog scale questionnaire | Up to 4 years
  Visual analog scale questionnaire regarding pain levels
Modified Japanese Orthopedic Association questionnaire (neck surgery only) | Up to 4 years
  Modified Japanese Orthopedic Association questionnaire regarding motor disfunction levels
Patient Satisfaction (neck surgery only) | Up to 4 years
  Patient satisfaction questionnaire regarding satisfaction of neck surgery
Scoliosis Research Society (SRS) 22r Survey | Up to 4 years
  Scoliosis Research Society (SRS) 22r Survey regarding pain, mental health, and function of the subject.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Christopher Kleck, MD, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Only aggregate data will be shared with the other investigators in the group